CLINICAL TRIAL: NCT05681117
Title: The Effect of Multi-Component Nutrition Education on Nutrition Health Literacy and Nutrition Attitudes of University Students
Brief Title: Increasing Nutritional Health Literacy With Multi-component Nutrition Education Given to University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BETÜL BAŞAR KARA (Other)
Responsible Party: Sponsor-Investigator, BETÜL BAŞAR KARA, lecturer, Bozok University
Organization: Bozok University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BOZOKU-NURSİNG-BBK-01
Record Dates: First submitted 2022-06-16; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Nutrition, Healthy
Keywords: University students; Nutrition Education; Nutrition Literacy

STUDY DESIGN:
Intervention Model Description: Randomized controlled (parallel group) experimental research design in the research pre-test-post-test order
Who Masked: Investigator, Outcomes Assessor
Masking Description: In order to eliminate bias, the data of the study were collected and recorded by an unbiased researcher (co-researcher) who did not know the researcher-trained groups. The statistics of the research were made by an independent statistician who did not know the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): No intervention will be made in the control group.
- Experimental group (Experimental): Class-based nutrition education, online intervention (SMS reminders with tips for healthy eating), distribution of brochures prepared in accordance with the educational content, and a controversial supermarket tour were organized in the experimental group as multiple interventions. Class-based nutrition education was given as a 40-minute session once a week for 4 weeks. Nutrition education content has been prepared as 4 modules in line with the current literature.
  Interventions: Other: multi-component nutrition education

INTERVENTIONS:
Other: multi-component nutrition education — Classroom-based nutrition education 40 minutes once a week for 4 weeks
  SMS Reminders SMS reminders containing healthy nutrition tips 2 times a week, 1 weekday, 1 weekend, starting with nutrition education and throughout the education (4 weeks)
  Brochure Distribution Brochures prepared in accordance with the content of classroom-based nutrition education were distributed immediately after the nutrition education.
  Controversial Supermarket Tour Nutrition label reading activity aimed at gaining the ability to evaluate product contents, in line with the information explained in module 4, in the supermarket tour planned to be organized once with an appropriate number of student groups (maximum 7 people) after the nutrition education
  Arms: Experimental group

SUMMARY:
In this study, based on the integrated health literacy model, it is aimed to increase the nutritional literacy level of university students and to strengthen their healthy nutritional attitudes with the multi-component nutrition education to be given.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of the multi-education initiative, organized according to the integrated health literacy model, on the nutritional health literacy and nutritional attitudes of university students.The research will be conducted with a randomized controlled (parallel group) experimental research design in the pre-test-post-test order.

The universe of the research; It consists of 1658 students who continue their education at Yozgat Bozok University Faculty of Education. All of the students in Bozok University Faculty of Education who volunteered to participate in the research were included in the study and a total of 1014 students were reached. The number of students who were suitable for the sample selection criteria (n:246) to be included in the experimental and control groups was determined by power analysis. In the power analysis, the sample size was calculated as at least 26 individuals for each group, with 95% confidence (1-α), 80% test power (1-β) and d=0.8 effect size (taking large effect width). Since it is thought that there may be data losses, 15% more of this number (n:32 for each group) was taken. The data of the study were collected with Personal Information Form, Adult Nutrition Literacy Assessment Tool, and Attitude towards Healthy Eating Scale. After obtaining the voluntary consent form from the students with low nutritional literacy level and who agreed to participate in the study, they would be blocked according to gender and then randomly assigned as 32 participants as experimental group and 32 as control group.

Control Group:

No intervention will be made in the control group. When the application part of the thesis is finished, handbooks about nutrition prepared by the researcher will be distributed to this group.

Experimental Group:

As multiple interventions, classroom-based nutrition education, online intervention (SMS reminders with healthy eating tips), brochures prepared in accordance with the educational content, and a controversial supermarket tour were made to the experimental group as multiple interventions.

Class-based nutrition education was given in 40-minute sessions once a week for 4 weeks.Multi-component nutrition education contents were prepared in accordance with the current literature and presented to the opinion of experts (Three Public Health Nursing Faculty Members, Three Nutrition and Dietetics Faculty Members, Three Educational Sciences Faculty Members and Two Clinical Dieticians) and their evaluations were taken in terms of content with the expert opinion form.

Class-based nutrition education has been prepared as 4 modules. Module 1: basic nutritional information and reliable resources Module 2: Healthy Eating Module 3: Evaluating information about nutrition Module 4: Reading Food Labels The prepared content was presented to the expert board and its evaluations were taken in terms of content. Methods used in education; Presentation (transfer information, question and answer, discussion), brainstorming, concept map method, fishbone method, case discussion and demonstration (show and make).

SMS Reminders:

Starting with the nutrition education, SMS reminders containing healthy nutrition tips were sent twice a week, once a week, and twice a week, once a week, during the education (4 weeks).

Brochure Distribution:

Brochures prepared in accordance with the content of classroom-based nutrition education were distributed immediately after the nutrition education.

Controversial Supermarket Tour:

Participants who completed the classroom-based nutrition education were divided into four groups (7 people in each group). The researcher organized a controversial supermarket tour for each group separately and each tour lasted an average of 45 minutes. In order to encourage participation in the controversial supermarket tour, gift vouchers were prepared for the students to use in the same supermarket and distributed to the students after the tour. In line with the information explained in the fourth module, which is the nutrition label reading module, a food label reading activity was carried out to gain the ability to evaluate the product contents. Before this activity, the controversial supermarket tour guideline was prepared by the researcher and the tour was conducted within the scope of this guideline. In the application of food label reading, labels were determined, especially unhealthy industrial products and one product from each food group. When it comes to the aisles of the determined products, these products were distributed to all students and the students were asked to evaluate the content of the label. The missing important points were emphasized by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of Yozgat Bozok University Faculty of Education
* Volunteering to participate in the research
* According to the Adult Nutrition Literacy Assessment Tool scale; Being at the level of nutritional literacy between 0-11 points inadequate, 12-23 points at the border.

Exclusion Criteria:

* According to the Adult Nutrition Literacy Assessment Tool scale; Adequate nutrition literacy level between 24-35 points
* living with family
* Having a chronic disease (diabetes, hypertension, hyperthyroidism, anemia, osteoporosis, celiac, etc. digestive system diseases)
* Being a foreign student

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Adult Nutrition Literacy Assessment Tool (YBOYDA) | 1 year
  The four-choice multiple-choice scale consists of 28 questions and 5 subsections.
  It is classified as insufficient nutrition literacy level between 0-11 points, borderline between 12-23 points and adequate nutrition literacy level between 24-35 points over the total score.

SECONDARY OUTCOMES:
Personal Information Form | 1 year
  The personal information form was prepared by the researcher in accordance with the proximal (near) and distal (far) determinants of the Integrated SFM model.
  The first part of the form consists of individual determinants (age, gender, race, socioeconomic status, education, occupation, employment, income) and situational determinants (social support, family and peer influence, media, physical environment), which are the proximal determinants of the model.
  The second part of the form consists of social and environmental determinants (demographic situation, culture, language, political forces, social systems), which are the distal determinants of the model. The personal information form consists of 28 questions in total.
Attitude Scale Towards Healthy Eating (SBIÖ) | 1 year
  SIBS has a structure consisting of 21 items and 4 factors. These factors were named as Knowledge About Nutrition (KHB), Emotion Towards Nutrition (BYD), Positive Nutrition (OB) and Malnutrition (BP).
  The lowest score that can be obtained from SBIÖ is 21, and the highest score is 105. It is explained that the participants from the SBIÖ have an attitude towards healthy eating with 21 points very low, 23-42 points low, 43-63 points medium, 64-84 points high, and 85-110 points ideally high.

CONTACTS AND LOCATIONS:
Overall Officials: bozok unıversity sağlık hizmetleri, Principal Investigator — www.bozok.edu.tr
Locations (1):
- Bozok Unıversity, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No